CLINICAL TRIAL: NCT01604356
Title: Acupuncture for the Treatment of Vision Loss Due to Retinitis Pigmentosa
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Ava Bittner, Principal Investigator, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00050691
Record Dates: First submitted 2012-05-21; First posted 2012-05-23 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Retinitis Pigmentosa
Keywords: retinitis pigmentosa
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electro-acupuncture (Experimental)
  Interventions: Procedure: Electro-acupuncture

INTERVENTIONS:
Procedure: Electro-acupuncture — Ten treatment sessions at our center during a two week period (5 sessions per week). Each session will last approximately 30 minutes. The intervention will involve the placement of acupuncture needles in a standard set of points across all patients, located on the head, around the eyes, on the abdomen, on the hands, feet, arms and legs. An electro-acupuncture device [Transcutaneous electrical nerve stimulator (TENS) unit by Lhasa OMS Inc.; model AWQ-104L] and will be used on four of the acupuncture points (two per session) located on the forehead, and side of the face/temple.

SUMMARY:
Retinitis Pigmentosa (RP) patients are interested in trying alternative therapies to attempt to slow, halt or reverse the retinal disease process, and claim success with some approaches such as acupuncture, but this potential treatment has not been put to the test of objective, rigorous scientific study conducted in western society. In this pilot study, the investigators aim to evaluate an acupuncture treatment tailored to the RP population for its feasibility to improve visual function, specifically visual field and dark adaptation. The study results may provide a basis for eye care providers' recommendations to RP patients regarding whether to consider acupuncture as a potential treatment modality. If our hypotheses regarding improvements in vision beyond typical test variability are supported, our future research goals include the conduct of a larger clinical trial with involving randomization and a placebo control for acupuncture in RP.

ELIGIBILITY:
Inclusion Criteria:

* Age 10+
* Diagnosis of retinitis pigmentosa
* Best-corrected visual acuity better than 20/400 in at least one eye
* More than 20% loss of Goldmann Visual Field area (III4e) in at least one eye
* Able and willing to participate in all study visits in Baltimore for the 8-week program
* Provide informed consent

Exclusion Criteria:

* Very severe vision losses in both eyes (e.g., hand motions or light perception only) with difficulty performing the proposed vision tests
* Vision loss due to ocular diseases other than RP, cystoid macular edema, or cataracts
* Schedules do not permit participation in all study visits
* Previous acupuncture treatment in the last 6 months
* Inability to understand study procedures or communicate responses to visual stimuli in a consistent manner (cognitive impairment)
* Dementia; Long or short-term memory loss
* Unable to read or speak English
* Smoking, substance abuse, or illegal drug use
* Receiving current psychiatric care (i.e. unstable emotional and mental health status)
* History of excessive bleeding

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Dark-adapted (Scotopic) Full-field Stimulus Test | initial response within 2 weeks after completion of treatment

SECONDARY OUTCOMES:
Goldmann visual fields | initial response within 2 weeks of treatment completion
PC-based vision tests (visual acuity, contrast sensitivity, visual field) | initial response within 2 weeks of treatment completion
ETDRS visual acuity | initial response within 2 weeks of treatment completion
Pelli-Robson contrast sensitivity | initial response within 2 weeks of treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States